CLINICAL TRIAL: NCT06288607
Title: Safety and Efficacy of High-Intensity Macrofocused Ultrasound for Solar Lentigo in Chinese Population: A Prospective Study
Brief Title: Safety and Efficacy of High-Intensity Macrofocused Ultrasound for Solar Lentigo in Chinese Population
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-708
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Solar Lentigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with solar lentigo
  Interventions: Device: High intensity focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China)

INTERVENTIONS:
Device: High intensity focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China) — Before treatment, a 2-3mm thick medical condensation gel is evenly applied on the face. Patients are to be treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Following the treatment, local cooling with an ice pack was performed for 10 min to reduce redness and swelling. Patients were followed up at 2, 4, 6, and 8 weeks. Clinical images and non-invasive skin assessments were collected at baseline and during each visit.

SUMMARY:
This trial is a single-center, prospective study. The study proposes to recruit 20 patients with solar lentigo on both sides of the face. Patients are to be treated with high-intensity focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China). oth sides of the face received treatment with identical parameters. The facial images are collected with dermoscope (DermLite DL4,3 Gen Inc., San Juan Capistrano, CA, USA), VISIA® (Canfield Company, USA) and a two-photon microscope (Transcend Vivoscope, China). For dermoscopy images, ImageJ software was then utilized to perform Lab* conversion on both the lesional area and the surrounding non-lesional areas. Measurements of transepidermal water loss (TEWL) values, skin elasticity and related images at the same location, along with adverse events, physician and subjective global aesthetic improvement scale scores are recorded before and at week2, week 4, week6 and week8.

ELIGIBILITY:
Inclusion Criteria:

1. adults between 18 and 70 years old, regardless of gender;
2. comply the clinical diagnostic criteria for solar lentigo on both sides of the face;
3. patients understand and are willing to participate in this clinical trial and voluntarily sign an informed consent form;

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or who plan to become pregnant during the trial period;
2. those who are allergic to medical condensation gel;
3. those with photosensitive diseases, immune deficiencies, or those who are taking immunosuppressants;
4. those with scar physique;
5. those with inflammatory or infectious skin diseases;
6. those who have systemically used retinoic acid in the last six months or topically applied retinoic acid drugs in the last three months, or have a history of sun exposure in the four weeks prior to treatment;
7. those who have undergone high-intensity focused ultrasound treatment within the last six months;

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population for this trial consisted of adult males and females, aged 18 to 70 years, diagnosed with solar lentigo. The participants were recruited from The First Affiliated Hospital with Nanjing Medical University.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants were to receive high intensity macro-focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China). No grouping was performed, both sides of the face received treatment with identical parameters. Before treatment, a 2-3mm thick medical condensation gel is evenly applied on the face. Patients are to be treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Following the treatment, local cooling with an ice pack was performed for 10 min to reduce redness and swelling. Patients were followed up at 2, 4, 6, and 8 weeks. Clinical images and non-invasive skin assessments were collected at baseline and during each visit. Outcomes were compared with data before and after treatment.
Period: Overall Study
Arm/Group | All Study Participants
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline population for this clinical trial consists of all enrolled participants. Baseline data were collected at the individual participant level and include the following characteristics: age, sex, race, Fitzpatrick Skin Type. These baseline data were collected for the entire participant group and represent the overall participant characteristics. The baseline data have been presented at the participant level.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 21
Fitzpatrick skin type [Count of Participants; unit: Participants] — The participants were categorized into one of the following six skin types:
  Type I: Very fair skin, always burns, never tans. Type II: Fair skin, burns easily, tans minimally. Type III: Medium skin, sometimes burns, gradually tans to light brown. Type IV: Olive skin, rarely burns, tans to a moderate brown. Type V: Brown skin, very rarely burns, tans to dark brown. Type VI: Dark brown or black skin, never burns, deeply pigmented. Generally, individuals with Type I-II skin are more susceptible to burning and may experience faster pigmentation changes in response to treatment.
  Participants
    Type I | 0
    Type II | 0
    Type Ⅲ | 15
    Type Ⅳ | 6
    Type V | 0
    Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Lab* Values of Lesional Area Using Dermoscopy and ImageJ
Description: Before treatment, one point on each side of every patient was selected for measurement. Follow-up measurements were taken at the same locations after treatment, and comparisons were made between the pre- and post-treatment values on the same side. This outcome measure involves the assessment of lesional areas in dermoscopy images, with the Lab* conversion of pigmentation intensity performed using ImageJ software. L* represents the lightness (brightness) of the lesion, where higher L* values indicate lighter lesions (improvement), ranging from 0 to 100. a* and b* represent the chromatic components (red-green and yellow-blue), both ranging from -128 to +127. Lower values in these components indicate lighter pigmentation, while higher values suggest darker lesions.
Time Frame: week0, week2, week4, week6 and week8
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- All Study Participants: All participants were to receive high intensity macro-focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China). Both sides of the face received treatment with identical parameters. Before treatment, a 2-3mm thick medical condensation gel is evenly applied on the face. Patients are to be treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Following the treatment, local cooling with an ice pack was performed for 10 min to reduce redness and swelling. Patients were followed up at 2, 4, 6, and 8 weeks. Clinical images and non-invasive skin assessments were collected at baseline and during each visit. Each area was treated first at 3.0mm then at 4.5mm depth. Since the individual effects of each depth could not be determined during follow-up, the results reflect the combined effects of both depths.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
unitless
  L* of left side at baseline | 68.850 (5.952)
  L* of left side at week2 | 72.103 (8.324)
  L* of left side at week4 | 73.147 (6.483)
  L* of left side at week6 | 72.633 (5.007)
  L* of left side at week8 | 73.646 (3.532)
  L* of right side at baseline | 68.671 (8.038)
  L* of right side at week2 | 71.433 (8.643)
  L* of right side at week4 | 72.756 (7.085)
  L* of right side at week6 | 72.902 (4.843)
  L* of right side at week8 | 72.600 (5.285)
  a* of left side at baseline | 13.597 (5.582)
  a* of left side at week2 | 11.476 (5.690)
  a* of left side at week4 | 9.948 (3.420)
  a* of left side at week6 | 9.787 (3.633)
  a* of left side at week8 | 9.295 (2.826)
  a* of right side at baseline | 13.099 (6.385)
  a* of right side at week2 | 11.818 (6.368)
  a* of right side at week4 | 10.065 (4.108)
  a* of right side at week6 | 9.732 (2.830)
  a* of right side at week8 | 9.233 (2.969)
  b* of left side at baseline | 18.324 (8.494)
  b* of left side at week2 | 12.285 (6.681)
  b* of left side at week4 | 12.464 (7.880)
  b* of left side at week6 | 10.642 (4.954)
  b* of left side at week8 | 11.482 (6.779)
  b* of right side at baseline | 17.592 (7.356)
  b* of right side at week2 | 14.036 (5.686)
  b* of right side at week4 | 12.348 (7.172)
  b* of right side at week6 | 11.687 (4.498)
  b* of right side at week8 | 12.737 (4.198)

2. Primary Outcome: Physician Global Aesthetic Improvement Scale Score
Description: Two physicians independently assessed the overall unilateral condition of each patient at various follow-up time points after treatment, comparing the numerical values obtained after treatment for the same side. Both scores were averaged as the final data. The Physician Global Aesthetic Improvement Scale (PGAIS) is a 5-point scale used to rate the global aesthetic improvement in appearance compared to pretreatment, as judged by the investigator. The scale ranges from -1 (worsening) to 3 (very much improved). The higher score indicates the better improving effect.
Time Frame: week2, week4, week6 and week8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Study Participants: All participants were to receive high intensity macro-focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China). No grouping was performed, both sides of the face received treatment with identical parameters. Before treatment, a 2-3mm thick medical condensation gel is evenly applied on the face. Patients are to be treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Following the treatment, local cooling with an ice pack was performed for 10 min to reduce redness and swelling. Patients were followed up at 2, 4, 6, and 8 weeks. Clinical images and non-invasive skin assessments were collected at baseline and during each visit. Outcomes were compared with data before and after treatment. Each area was treated first at 3.0mm then at 4.5mm depth. Since the individual effects of each depth could not be determined during follow-up, the results reflect the combined effects of both depths.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
score on a scale
  scores of left side at week2 | 0.800 (0.510)
  scores of left side at week4 | 1.368 (0.470)
  scores of left side at week6 | 1.850 (0.477)
  scores of left side at week8 | 1.889 (0.624)
  scores of right side at week2 | 0.900 (0.436)
  scores of right side at week4 | 1.263 (0.620)
  scores of right side at week6 | 1.850 (0.572)
  scores of right side at week8 | 1.944 (0.589)

3. Primary Outcome: Subjective Global Aesthetic Improvement Scale Score
Description: At each follow-up time point after treatment, patients self-evaluated their unilateral overall condition and compared the numerical values of the same side before and after treatment. This process was repeated at every follow-up time point. The Subjective Global Aesthetic Improvement Scale (SGAIS) is a 5-point scale used to rate the global aesthetic improvement in appearance compared to pretreatment, as judged by the patients. The scale ranges from -1 (worsening) to 3 (very much improved). The higher score indicates the better improving effect.
Time Frame: week2, week4, week6 and week8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
score on a scale
  scores of left side at week2 | 1.211 (0.979)
  scores of left side at week4 | 1.619 (0.669)
  scores of left side at week6 | 2.050 (0.589)
  scores of left side at week8 | 1.833 (0.725)
  scores of right side at week2 | 1.158 (0.962)
  scores of right side at week4 | 1.667 (0.796)
  scores of right side at week6 | 2.000 (0.632)
  scores of right side at week8 | 1.833 (0.725)

4. Primary Outcome: Transepidermal Water Loss (TEWL) Measurement of Lesional Area
Description: Before treatment, one point on each side of every patient was selected for measurement. Follow-up measurements were taken at the same locations after treatment, and comparisons were made between the pre- and post-treatment values on the same side. Transepidermal Water Loss (TEWL) TEWL can be used to assess a patient's skin barrier function, with lower values indicating stronger barrier function.
  This outcome measure involves the assessment of Transepidermal Water Loss (TEWL), which quantifies the amount of water evaporating through the skin. TEWL is a key indicator of skin barrier function and hydration levels. In this study, TEWL was measured using Tewameter Hex (Courage Khazaka Electronic GmbH) that records the rate of water loss through the skin in g/m²/h (grams per square meter per hour). Lower TEWL values (less water loss) suggest an improved skin barrier, which is typically the result of effective treatment and increased skin hydration.
Time Frame: week0, week2, week4, week6 and week8
Measure: Mean (Standard Deviation); unit: g/m²/h
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
g/m²/h
  values of left side at baseline | 15.720 (4.715)
  values of left side at week2 | 15.097 (4.600)
  values of left side at week4 | 15.516 (4.820)
  values of left side at week6 | 14.042 (5.067)
  values of left side at week8 | 12.688 (3.927)
  values of right side at baseline | 14.834 (3.691)
  values of right side at week2 | 15.933 (3.934)
  values of right side at week4 | 16.136 (4.113)
  values of right side at week6 | 14.891 (3.848)
  values of right side at week8 | 13.478 (3.624)

5. Primary Outcome: Skin Elasticity Measurement of Lesional Area
Description: Before treatment, one point on each side of every patient was selected for measurement. Follow-up measurements were taken at the same locations after treatment, and comparisons were made between the pre- and post-treatment values on the same side. Skin elasticity was assessed using Cutometer Dual MPA580 (Courage Khazaka Electronic GmbH, Köln, Germany), which measures the skin's resistance to deformation and recovery after deformation. The R-value represents the ratio of skin's ability to resist deformation (stiffness) and its ability to return to its original shape (elasticity). Higher R-values (greater elasticity) suggest that the skin is more resilient and can return to its original shape after deformation, indicating healthy skin with good elasticity and tone.
Time Frame: week0, week2, week4, week6 and week8
Measure: Mean (Standard Deviation); unit: dimensionless unit
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
dimensionless unit
  values of left side at baseline | 0.710 (0.126)
  values of left side at week2 | 0.744 (0.127)
  values of left side at week4 | 0.810 (0.106)
  values of left side at week6 | 0.792 (0.101)
  values of left side at week8 | 0.825 (0.073)
  values of right side at baseline | 0.736 (0.142)
  values of right side at week2 | 0.752 (0.126)
  values of right side at week4 | 0.783 (0.125)
  values of right side at week6 | 0.821 (0.104)
  values of right side at week8 | 0.807 (0.066)

ADVERSE EVENTS:
Time Frame: 2 weeks, 4 weeks, 6 weeks and 8 weeks
Description: Patients were treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Given that each patient was subjected to treatment with both 3.0mm and 4.5mm handpieces, it was not possible to distinguish adverse events related to different depths during follow-up. Therefore, these events were synthesized into an overall assessment of adverse events.
Groups:
- Patients: Patients with solar lentigo
  All participants were to receive high intensity macro-focused ultrasound (MFUS One, Hunan Peninsula Medical Technology Co., Ltd., China). No grouping was performed, both sides of the face received treatment with identical parameters. Before treatment, a 2-3mm thick medical condensation gel is evenly applied on the face. Patients are to be treated with two macro-focused handpieces with focal depths at 3.0 mm (D3.0) and 4.5 mm (D4.5) on both side. Following the treatment, local cooling with an ice pack was performed for 10 min to reduce redness and swelling. Patients were followed up at 2, 4, 6, and 8 weeks. Clinical images and non-invasive skin assessments were collected at baseline and during each visit. Outcomes were compared with data before and after treatment.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients (N=21)
Pain sensation post treatment (Skin and subcutaneous tissue disorders) | 2
edema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT06288607/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT06288607/ICF_001.pdf